CLINICAL TRIAL: NCT00006246
Title: Phase I Study of Intrathecal Spartaject-Busulfan in Children With Neoplastic Meningitis
Brief Title: Busulfan in Treating Children and Adolescents With Refractory CNS Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James M. Boyett/PBTC Operations and Biostatistics Center Executive Director, Pediatric Brain Tumor Consortium
Purpose: Treatment
Other Study IDs: CDR0000068178; PBTC-004
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Brain and Central Nervous System Tumors; Childhood Germ Cell Tumor; Leukemia; Lymphoma; Metastatic Cancer; Retinoblastoma; Sarcoma
Keywords: recurrent childhood acute lymphoblastic leukemia; childhood infratentorial ependymoma; recurrent childhood rhabdomyosarcoma; recurrent childhood brain tumor; recurrent retinoblastoma; recurrent childhood lymphoblastic lymphoma; childhood central nervous system germ cell tumor; recurrent childhood acute myeloid leukemia; recurrent/refractory childhood Hodgkin lymphoma; leptomeningeal metastases; childhood high-grade cerebral astrocytoma; childhood oligodendroglioma; childhood choroid plexus tumor; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; recurrent childhood large cell lymphoma; recurrent childhood brain stem glioma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; recurrent childhood visual pathway and hypothalamic glioma; recurrent childhood ependymoma; recurrent childhood malignant germ cell tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Leukemia; Lymphoma; Neoplasm Metastasis; Retinoblastoma; Sarcoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Meningeal Carcinomatosis; Astrocytoma; Oligodendroglioma; Choroid Plexus Neoplasms; Dendritic Cell Sarcoma, Interdigitating; Medulloblastoma; Optic Nerve Glioma; Familial ependymoma | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: busulfan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the safety of delivering intrathecal busulfan in children and adolescents who have refractory CNS cancer and to estimate the maximum tolerated dose of this treatment regimen.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the qualitative and quantitative toxicities of intrathecally administered busulfan in children and adolescents with refractory CNS malignancies.
* Determine the maximum tolerated dose of this treatment regimen in these patients.
* Determine the cerebrospinal fluid and serum pharmacokinetics of this treatment regimen in these patients.
* Determine the efficacy of this treatment regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive intrathecal busulfan twice a week, at least 3 days apart, for 2 weeks. Patients with complete or partial response or stable disease may continue therapy once a week for 2 weeks, once a week every other week for 2 treatments, and then once a month thereafter in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of busulfan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities.

Patients are followed every 3 months for the first year, every 6 months for 4 years, and then annually for 5 years.

PROJECTED ACCRUAL: Approximately 18-24 patients will be accrued for this study over 18-38 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed CNS malignancy, including any of the following:

  * Primary malignant brain tumor refractory to standard therapy and metastatic to the cerebrospinal fluid (CSF) or leptomeningeal subarachnoid space
  * Recurrent or persistent leptomeningeal leukemia, lymphoma, or germ cell tumor refractory to conventional therapy

    * In second or greater relapse
    * CSF white blood count greater than 5 cells/mm3 with blasts on cytospin OR
    * Evidence of leptomeningeal tumor by MRI
* No concurrent bone marrow disease
* No obstruction or compartmentalization of CSF flow on CSF flow study

PATIENT CHARACTERISTICS:

Age:

* 3 to 21

Performance status:

* Lansky 50-100% (under 10 years)
* Karnofsky 50-100% (10 to 21 years)

Life expectancy:

* Greater than 8 weeks

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 75,000/mm^3

Hepatic:

* Bilirubin normal for age
* ALT and AST less than 5 times upper limit of normal (ULN)
* No hepatic disease

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Glomerular filtration rate greater than 70 mL/min
* No renal disease

Cardiovascular:

* No cardiac disease

Pulmonary:

* No pulmonary disease

Other:

* No uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas)
* At least 1 week since prior intrathecal chemotherapy (2 weeks for cytarabine) and recovered
* Evidence of subsequent disease progression
* Concurrent systemic chemotherapy allowed for recurrent disease after first course of treatment except for the following:

  * Chemotherapy targeted at leptomeningeal disease
  * Other phase I agent
  * Any agent that significantly penetrates the CSF (e.g., high dose methotrexate greater than 1 g/m2, thiotepa, high dose cytarabine, fluorouracil, IV mercaptopurine, nitrosoureas, or topotecan)
  * Any agent that causes serious unpredictable CNS side effects

Endocrine therapy:

* Prior dexamethasone allowed with decreasing or stable dose at least one week before study
* Concurrent dexamethasone or prednisone with chemotherapy regimen allowed

Radiotherapy:

* At least 1 week since prior focal irradiation to the brain or spine
* At least 8 weeks since prior craniospinal irradiation
* No concurrent cranial or craniospinal irradiation

Surgery:

* Not specified

Other:

* No other concurrent intrathecal or systemic therapy for leptomeningeal disease

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2000-11; Primary Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Toxicities of IT administered busulfan in children and adolescents with refractory CNS malignancies
Maximum tolerated dose of IT administered busulfan
Serum and CSF pharmacokinetics of IT administered busulfan

CONTACTS AND LOCATIONS:
Overall Officials: Sri Gururangan, MD, Study Chair — Duke University
Locations (8):
- United States (8):
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Result] Gururangan S, Petros WP, Poussaint TY, Hancock ML, Phillips PC, Friedman HS, Bomgaars L, Blaney SM, Kun LE, Boyett JM. Phase I trial of intrathecal spartaject busulfan in children with neoplastic meningitis: a Pediatric Brain Tumor Consortium Study (PBTC-004). Clin Cancer Res. 2006 Mar 1;12(5):1540-6. doi: 10.1158/1078-0432.CCR-05-2094. PMID 16533779